CLINICAL TRIAL: NCT02137070
Title: Obesity and Type 2 Diabetes, Bariatric Surgery Effects on Brain Function
Brief Title: The WISE (Weightloss Intervention Surgical Effects) Brain Study
Acronym: WISEBrain
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201400034-N; 1R01DK099334-01A1 (NIH); OCR15981 (Other: Universiy of Florida)
Record Dates: First submitted 2014-05-09; First posted 2014-05-13 (Estimated); Results first posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-11

CONDITIONS: Diabetes; Weightloss
Keywords: Weightloss and brain function; Effects of bariatric surgery on brain function; Reduced glucose insulin changes and brain function
MeSH Terms: conditions — Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be retained for biomarker analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bariatric Surgery Candidates: Participants who are intending to have bariatric surgery for weight loss at local surgical centers or UFHEALTH & Shands Hospital.
  Interventions: Procedure: Bariatric Surgery Candidates
- Non surgical/Community volunteers: Healthy adults with body mass index >35 who will not undergo bariatric surgery for weight loss
  Interventions: Other: Non surgical/Community volunteers

INTERVENTIONS:
Procedure: Bariatric Surgery Candidates — Participants who are intending to have bariatric surgery for weight loss
  Groups: Bariatric Surgery Candidates
Other: Non surgical/Community volunteers — Healthy adults with body mass index >35 who will not undergo bariatric surgery for weight loss
  Groups: Non surgical/Community volunteers

SUMMARY:
This study is being done to learn about the changes that weight loss causes on brain function, memory and thinking ability in adults. The study does NOT cover any costs associated with bariatric surgery.

DETAILED DESCRIPTION:
There will be two groups of people studied:

One group has chosen (independently of this research study) to have weight loss surgery to help them lose weight.

Another group will not choose to have any weight loss surgery. All research participants will be tested on thinking and memory processes at the start of the study, after 12 weeks, and again at 18 months. They will have an MRI Brain Scan at those same times also to look at changes in the structure and function of the brain tissue.

Blood tests will be done to measure the sugar levels in the blood, and other proteins that may act as markers for disease.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index >35
* Diabetes or no diabetes
* Compatible with MRI Scanning
* Willing to give a small blood sample on 3 occasions
* Capable of providing informed consent

Exclusion Criteria:

* Prior neurological disorder
* Mini Mental Status Exam score
* Major psychiatric disturbance (schizophrenia, chronic intractable depression,
* Coronary revascularization, peripheral vascular disease
* Severe cardio vascular disease history
* Unstable medical conditions (cancer)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential bariatric surgery patients will have study specific information made available to them for their consideration at the bariatric or diabetes clinics at UFHealth & Shands Hospital, or at other community locations. Flyers will be posted in many community advertising locations in the North Florida region. Prospective participants must live in Gainesville, FL or the surrounding areas to be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2022-11 (Actual); Study Completion 2022-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald A Cohen, PHD, Principal Investigator — University of Florida
Locations (1):
- University of Florida - College of Public Health and Health Professions, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Fernando HJ, Cohen RA, Gullett JM, Friedman J, Ayzengart A, Porges E, Woods AJ, Gunstad J, Ochoa CM, Cusi K, Gonzalez-Louis R, Donahoo WT. Neurocognitive Deficits in a Cohort With Class 2 and Class 3 Obesity: Contributions of Type 2 Diabetes and Other Comorbidities. Obesity (Silver Spring). 2019 Jul;27(7):1099-1106. doi: 10.1002/oby.22508. Epub 2019 May 22. PMID 31116012

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bariatric Surgery Candidates | Non Surgical/Community Volunteers
Started | 150 | 47
Completed | 76 | 29
Not Completed | 74 | 18
Not completed — Adverse Event | 12 | 3
Not completed — Death | 2 | 0
Not completed — Lost to Follow-up | 24 | 9
Not completed — Physician Decision | 0 | 1
Not completed — Protocol Violation | 18 | 4
Not completed — Withdrawal by Subject | 18 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bariatric Surgery Candidates | Non Surgical/Community Volunteers | Total
Number analyzed (Participants) | 150 | 47 | 197
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 143 | 42 | 185
  >=65 years | 7 | 5 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.54 (11.51) | 52.29 (12.51) | 44.86 (12.44)
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean by intervention condition | 42.54 (11.51) | 52.29 (12.51) | 44.86 (12.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 32 | 150
  Male | 32 | 15 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 4 | 15
  Not Hispanic or Latino | 138 | 43 | 181
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 14 | 49
  White | 100 | 31 | 131
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 2 | 17
Region of Enrollment [Number; unit: participants]
  United States | 150 | 47 | 197
Age of study participants [Mean (Standard Deviation); unit: years] | 42.54 (11.51) | 52.29 (12.51) | 44.86 (12.44)

OUTCOME MEASURES:

1. Primary Outcome: Change in BOLD fMRI Signal
Description: Brain activation changes will change in the frontal cortex and hippocampus.
  * z-score is a transformation of the Pearson's (r) correlation coefficient of the BOLD timeseries between two brain regions
  * a value of < 0 suggests a weakening of the connections between brain areas; and a value of > 0 suggests a strengthening of the connections between brain areas
  * A value of r=0 indicates that two brain regions were functionally disconnected
Time Frame: Change from baseline at 18 months
Population: 37 individuals completed pre-surgery MRI at baseline and 18-month follow-up.
Measure: Mean (Standard Deviation); unit: Connectivity Fisher-z transformation
Arm/Group | Bariatric Surgery Candidates | Non Surgical/Community Volunteers
Number analyzed (Participants) | 20 | 17
Connectivity Fisher-z transformation
  Baseline - Seed (R Hippocampus) to cluster (MNI -44 -26 46) | 0.10 (0.10) | 0.08 (0.09)
  Follow-up - Seed (R Hippocampus) to cluster (MNI -44 -26 46) | 0.18 (0.13) | -0.01 (0.13)
  Baseline - Seed (L Hippocampus) to cluster (MNI 16, -24, 56) | 0.09 (0.09) | 0.09 (0.10)
  Follow-up - Seed (L Hippocampus) to cluster (MNI 16, -24, 56) | 0.16 (0.14) | -0.03 (0.14)
  Baseline - Seed (R Frontal Pole) to cluster (MNI 60, -26, 24) | 0.07 (0.09) | 0.10 (0.09)
  Follow-up - Seed (R Frontal Pole) to cluster (MNI 60, -26, 24) | 0.21 (0.16) | 0.03 (0.14)
  Baseline - Seed (L Frontal Pole) to cluster (MNI 60, 08, -30) | 0.05 (0.10) | 0.10 (0.07)
  Follow-up - Seed (L Frontal Pole) to cluster (MNI 60, 08, -30) | 0.16 (0.11) | 0.00 (0.10)
  Baseline - Seed (R Inferior Frontal Gyrus) to cluster (MNI -66, -24, -20) | 0.12 (0.09) | 0.15 (0.08)
  Follow-up - Seed (R Inferior Frontal Gyrus) to cluster (MNI -66, -24, -20) | 0.24 (0.09) | 0.09 (0.10)
  Baseline - Seed (R Inferior Frontal Gyrus) to cluster (MNI 40, -22, 52) | 0.22 (0.12) | 0.20 (0.10)
  Follow-up - Seed (R Inferior Frontal Gyrus) to cluster (MNI 40, -22, 52) | 0.34 (0.10) | 0.14 (0.12)
  Baseline - Seed (R Inferior Frontal Gyrus) to cluster (MNI 02, -38, 66) | 0.14 (0.12) | 0.12 (0.11)
  Follow-up - Seed (R Inferior Frontal Gyrus) to cluster (MNI 02, -38, 66) | 0.25 (0.13) | 0.06 (0.12)
  Baseline - Seed (L Inferior Frontal Gyrus) to cluster (MNI 32, 14, -16) | 0.12 (0.11) | 0.11 (0.09)
  Follow-up - Seed (L Inferior Frontal Gyrus) to cluster (MNI 32, 14, -16) | 0.22 (0.09) | 0.01 (0.10)
  Baseline - Seed (Anterior Cingulate) to cluster (MNI 60, -06, -04) | 0.07 (0.10) | 0.10 (0.10)
  Follow-up - Seed (Anterior Cingulate) to cluster (MNI 60, -06, -04) | 0.17 (0.10) | 0.00 (0.13)
Statistical Analysis 1: Comparison: Bariatric Surgery Candidates vs Non Surgical/Community Volunteers; Analysis of variance comparing change scores from 18 months post-surgery relative to pre-surgical baseline were performed. Change in the surgical group was compared to change for the non-surgical controls. The dependent measures were connectivity strengths seeding from the hippocampus and left dorsal lateral pre-frontal cortex to other cortical areas; Test type: Superiority; p < 0.01, 2x2 Factorial ANOVA in CONN — Voxel-size (p-FWE < 0.01) and voxel-peak (p-unc < 0.001) were corrected for multiple comparisons; 2x2 Factorial ANOVA in CONN - Group (Bariatric surgery vs. control) & time (pre-surgery baseline vs. 18-month follow-up)

ADVERSE EVENTS:
Time Frame: 18 months
Description: Consistent with clinicaltrials.gov
Groups:
- Surgical Group: Participants that received surgery
- Control Group: Participants that did not receive surgery
Arm/Group | Surgical Group | Control Group
All-Cause Mortality (participants affected / at risk) | 2/150 | 0/47
Serious Adverse Events (participants affected / at risk) | 5/150 | 0/47
Other Adverse Events (participants affected / at risk) | 11/150 | 3/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Surgical Group (N=150) | Control Group (N=47)
Post-surgical Symptoms (Gastrointestinal disorders) | 3 | 0
High BDI (Psychiatric disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Surgical Group (N=150) | Control Group (N=47)
MRI symptoms (General disorders) | 4 | 2
Blood draw problems (General disorders) | 3 | 1
Other tasks (General disorders) | 1 | 0
Survey Questions/Cognitive questions (Social circumstances) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol: Protocol Document (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT02137070/Prot_000.pdf
  • Study Protocol and Informed Consent Form: ICF Document (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT02137070/Prot_ICF_001.pdf